CLINICAL TRIAL: NCT04401202
Title: Effects of Nigella Sativa as a Treatment of Patients With Upper Respiratory Tract Infection Caused by SARS-coronavirus-2: a Prospective, Randomized, Open-label, Controlled Clinical Study
Brief Title: Nigella Sativa in COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Dr Abdulrahman E. Koshak, Assistant Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 266-20
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19; SARS-CoV-2; Nigella sativa; Herbal
MeSH Terms: conditions — COVID-19 | interventions — Nigella sativa oil

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label, controlled clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSO (Experimental): Nigella sativa oil 500mg softgel capsules in oral twice daily dose for 10 days
  Interventions: Dietary Supplement: Nigella sativa oil
- Control (No Intervention): Standard of care

INTERVENTIONS:
Dietary Supplement: Nigella sativa oil — Nigella sativa oil 500mg softgel capsules in oral twice daily dose for 10 days
  Arms: NSO

SUMMARY:
Natural products with immunomodulation and antiviral activity showed a promising improvement in the outcomes of some viral infectious diseases both in preclinical and primitive clinical studies. The aim of this study is to utilize Saudi FDA licensed Nigella sativa (NS) seed oil towards improving disease outcomes in adult patients diagnosed with mild COVID-19. The study will be a prospective, open-label, non-randomized controlled pilot trial. Patients will be supplemented (add-on) with one capsule of black seed oil twice daily for 10 days. The primary outcome will be the proportion of patients who clinically recovered on day 14. The secondary outcomes will be clinical parameters and routine laboratory tests. If encouraging outcomes occurred, NS supplementation may be recommended as an add-on to standard care protocol to enhance the recovery from COVID-19 disease in the current emerging situation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild COVID19 upper respiratory tract infection and with no evidence of pneumonia
* Adult (18 Years and above)
* Written informed consent prior to initiation of any study procedures by the patient (or legally authorized representative).
* Understands and agrees to comply with planned study procedures.
* Has laboratory-confirmed novel coronavirus (SARS-CoV-2) infection as determined by polymerase chain reaction (PCR) available at KAUH.

Exclusion Criteria:

* Patients with pneumonia or severe illness requiring admission to ICU.
* Severe chronic kidney disease (i.e. estimated glomerular filtration rate (eGFR) < 30) or end stage renal disease requiring dialysis
* Sever chronic liver disease (Alanine transaminase/aspartate transaminase (ALT/AST) > 5 times the upper limit of normal).
* Pregnancy or breast feeding.
* Anticipated transfer to another hospital which is not a study site within 72 hours.
* Allergy to any study medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koshak AE, Koshak EA, Mobeireek AF, Badawi MA, Wali SO, Malibary HM, Atwah AF, Alhamdan MM, Almalki RA, Madani TA. Nigella sativa for the treatment of COVID-19: An open-label randomized controlled clinical trial. Complement Ther Med. 2021 Sep;61:102769. doi: 10.1016/j.ctim.2021.102769. Epub 2021 Aug 15. PMID 34407441
- [Derived] Koshak AE, Koshak EA, Mobeireek AF, Badawi MA, Wali SO, Malibary HM, Atwah AF, Alhamdan MM, Almalki RA, Madani TA. Nigella sativa supplementation to treat symptomatic mild COVID-19: A structured summary of a protocol for a randomised, controlled, clinical trial. Trials. 2020 Aug 8;21(1):703. doi: 10.1186/s13063-020-04647-x. PMID 32771034

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 233 cases assessed for eligibility. 50 cases were excluded because; Asymptomatic (31), Pregnant (3), Declined to participate (n= 7), Failed communication (n= 9)
Period: Overall Study
Arm/Group | Control | Nigella Sativa Oil
Started | 92 | 91
Completed | 86 | 87
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Hospitalized | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nigella Sativa Oil | Control | Total
Number analyzed (Participants) | 87 | 86 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10) | 35 (11) | 35 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 80
  Male | 46 | 47 | 93
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (6.1) | 27.2 (5.5) | 27.1 (5.7)
Smoker [Count of Participants; unit: Participants] | 12 | 9 | 21
Pre-enrollment days [Mean (Standard Deviation); unit: days] — The time from the first day of symptoms until the day of enrollment
  days | 3.5 (2.1) | 4 (3.1) | 3.7 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Recovery Within 14 Days After Randomization
Description: The Percentage of patients who had clinical recovery within 14 days after randomization (clinical recovery was defined as three days of no symptoms)
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Nigella Sativa Oil | Control
Number analyzed (Participants) | 87 | 86
Participants | 54 | 31
Statistical Analysis 1: Comparison: Nigella Sativa Oil vs Control; Test type: Superiority; p = 0.001, Chi-squared

2. Secondary Outcome: The Number of Days to Recovery
Description: The number of days to recovery (number of symptomatic days)
Time Frame: Day 14
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nigella Sativa Oil | Control
Number analyzed (Participants) | 87 | 86
days | 11 [8 to 14] | 14 [11 to 14]

3. Secondary Outcome: Duration of Each Symptom
Description: Duration of each symptom in days
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nigella Sativa Oil | Control
Number analyzed (Participants) | 87 | 86
days
  Anosmia | 8.5 (3.9) | 10.4 (3.6)
  Runny nose | 2.5 (1.6) | 3.7 (2.5)
  Loss of appetite | 3.5 (2.9) | 5.5 (3.1)
  Chills | 2.1 (1) | 4.9 (3.4)

4. Secondary Outcome: Side Effects
Description: Side effects from the investigational treatment
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Nigella Sativa Oil | Control
Number analyzed (Participants) | 87 | 86
Participants | 3 | 0

5. Secondary Outcome: Hospital Admission Due to Disease Complications
Description: High severity of COVID-19 (mild cases does not require hospitalization)
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Nigella Sativa Oil | Control
Number analyzed (Participants) | 87 | 86
Participants | 0 | 4

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Nigella Sativa Oil | Control
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/86
Other Adverse Events (participants affected / at risk) | 3/87 | 0/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nigella Sativa Oil (N=87) | Control (N=86)
Gastrointestinal symptoms (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT04401202/Prot_SAP_000.pdf